CLINICAL TRIAL: NCT03205202
Title: Cataract and AMD in a Trial of a Multivitamin and Cocoa Extract (COSMOS-Eye)
Brief Title: Cataract and AMD in a Trial of a Multivitamin and Cocoa Extract
Acronym: COSMOS-Eye
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, William G. Christen, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2016P001612
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Cataract; Age Related Macular Degeneration
MeSH Terms: conditions — Cataract; Macular Degeneration | interventions — Chocolate; Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cocoa extract + multivitamin (Active Comparator): Dietary Supplement: Cocoa extract (2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin, and 50 mg theobromine)
  Dietary Supplement: Multivitamin
  Interventions: Dietary Supplement: Cocoa extract; Dietary Supplement: Multivitamin
- Cocoa extract + multivitamin placebo (Active Comparator): Dietary Supplement: Cocoa extract (2 capsules each day containing a total of 500 mg cocoa flavanols, including 80 mg (-)-epicatechin, and 50 mg theobromine)
  Dietary Supplement: Multivitamin placebo
  Interventions: Dietary Supplement: Cocoa extract; Dietary Supplement: Multivitamin placebo
- Cocoa extract placebo + multivitamin (Active Comparator): Dietary Supplement: Multivitamin
  Dietary Supplement: Cocoa extract placebo
  Interventions: Dietary Supplement: Multivitamin; Dietary Supplement: Cocoa extract placebo
- Cocoa extract placebo + multivitamin placebo (Placebo Comparator): Dietary Supplement: Cocoa extract placebo
  Dietary Supplement: Multivitamin placebo
  Interventions: Dietary Supplement: Cocoa extract placebo; Dietary Supplement: Multivitamin placebo

INTERVENTIONS:
Dietary Supplement: Cocoa extract
  Arms: Cocoa extract + multivitamin; Cocoa extract + multivitamin placebo
Dietary Supplement: Multivitamin
  Arms: Cocoa extract + multivitamin; Cocoa extract placebo + multivitamin
Dietary Supplement: Cocoa extract placebo
  Arms: Cocoa extract placebo + multivitamin; Cocoa extract placebo + multivitamin placebo
Dietary Supplement: Multivitamin placebo
  Arms: Cocoa extract + multivitamin placebo; Cocoa extract placebo + multivitamin placebo

SUMMARY:
COSMOS-Eye is an ancillary study of the COcoa-Supplement and Multivitamins Outcomes Study (COSMOS; NCT02422745). COSMOS is a randomized clinical trial of cocoa extract supplement (containing a total of 500 mg/d flavanols, including 80 mg (-)-epicatechins), and a standard multivitamin supplement to reduce the risk of cardiovascular disease and cancer among men aged 60 years and older and women aged 65 years and older. This ancillary study is being conducted among participants in COSMOS and will examine whether the cocoa extract supplement or the multivitamin supplement reduces the risk of cataract and AMD, two leading causes of visual impairment in US men and women.

DETAILED DESCRIPTION:
COSMOS-Eye is an ancillary study of cataract and AMD utilizing resources and data from the COcoa-Supplement and Multivitamins Outcomes Study (COSMOS), a randomized, double-blind, placebo-controlled, 2x2 factorial trial of a high-quality cocoa extract supplement (Mars Symbioscience) and Centrum Silver multivitamin (Pfizer) in the prevention of cardiovascular disease and cancer among 12,000 women aged ≥65 years and 6,000 men aged ≥60 years.

Women will be recruited among active Women's Health Initiative (WHI) Extension Study participants, and men will be recruited among non-randomized respondents to the VITamin D and OmegA-3 Trial (VITAL). Women who responded but were not randomized into VITAL will also be included as well as other women and men who express interest in research being conducted at Brigham and Women's Hospital.

Participants will take three pills each day: two capsules that contain either cocoa extract or cocoa extract placebo, and one tablet that contains either multivitamin or multivitamin placebo. Participants will receive their study pills in convenient calendar packs via U.S. mail.

Participants also will be asked to complete short mailed questionnaires each year. The questionnaires ask about health; lifestyle habits, such as diet, physical activity, and smoking; use of medications and dietary supplements; family history of illness and new medical diagnoses including cataract and AMD.

Participants who report cataract or AMD will be asked to provide contact information for their eye doctor(s) as well as written consent to obtain the medical records. Eye doctors will be contacted by mail and asked to complete a cataract (or AMD) questionnaire or, alternatively, forward a complete copy of the patient's medical records pertaining to the diagnosis.

After the COSMOS trial began, an advanced method to analyze cocoa flavanols was accredited by AOAC International as a First Action Official Method of Analysis https://doi.org/10.1093/jaoacint/qsaa132). This updated method relies on a reference material (RM8403) recently standardized and made commercially available by the U.S. National Institute of Standards and Technology. While the actual cocoa flavanol content of the COSMOS intervention remained unchanged throughout the trial, the application of this new analytical method led to expected changes in how the total cocoa flavanol content is now reported. Applying AOAC 2020.05/RM8403 to the COSMOS intervention, the total cocoa flavanol content of the COSMOS intervention is now 500 mg/day. Reporting of (-)-epicatechin content remained unaffected. Going forward, we will therefore apply AOAC 2020.05/RM8403 and report that the COSMOS intervention tested 500 mg/day of cocoa flavanols, including 80 mg of (-)-epicatechin.

ELIGIBILITY:
Participants in COSMOS who 1) report a diagnosis of cataract or AMD, or extraction of cataract, and 2) provide written consent to obtain the medical records for the reported endpoint, are eligible for this ancillary study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21442 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Cataract | 5 years
  Incident age-related cataract responsible for a reduction in best-corrected visual acuity to 20/30 or worse
Total AMD events | 5 years
  Composite of incident AMD plus cases of progression to advanced AMD (neovascular AMD plus central geographic atrophy) among participants with prevalent AMD at baseline

SECONDARY OUTCOMES:
Cataract surgery | 5 years
  Incident extraction of an age-related lens opacity
Total cataract events | 5 years
  Composite of incident cataract plus cataract surgery among participants with prevalent cataract at baseline
AMD | 5 years
  Incident AMD with or without vision loss
Visually-significant AMD | 5 years
  Incident AMD responsible for a reduction in best-corrected visual acuity to 20/30 or worse
Advanced AMD | 5 years
  Incident advanced AMD (neovascular or geographic atrophy)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christen WG, Rist PM, Moorthy MV, Smith DC, Holman B, Clar A, Glynn RJ, Mares JA, Sobrin L, Shadyab AH, Allison MA, Millen AE, Manson JE, Sesso HD; COSMOS Research Group. Cocoa Flavanol Supplementation and Risk of Age-Related Macular Degeneration: An Ancillary Study of the COSMOS Randomized Clinical Trial. JAMA Ophthalmol. 2025 May 1;143(5):429-437. doi: 10.1001/jamaophthalmol.2025.0353. PMID 40146119